CLINICAL TRIAL: NCT07303933
Title: The Association Between Head Cooling and Cognition, Neuroinflammatory Cytokines, Menstrual Cycle, Sleep Patterns, Mental Health and Concussions
Brief Title: Female Concussion Head Cooling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Owen Griffith, Assistant Teaching Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Female Concussion Head Cooling
Record Dates: First submitted 2025-12-20; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Concussion (Diagnosis); Concussion Post Syndrome; Concussion, Mild
Keywords: Brain cooling; Concussion; Neuroinflammation; Mental Health; Cognition; Menstrual cycle; Female
MeSH Terms: conditions — Brain Concussion; Disease; Post-Concussion Syndrome; Neuroinflammatory Diseases; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This will be a straight forward parallel intervention model. Even numbers of participants will be randomly assigned to the treatment or control arms. The treatment group will receive the brain cooling intervention during their visits (on top of normal clinical care), while the control group will receive their normal clinical care. All other environmental, timing, and testing measures will remain constant between the groups as indicated in the study description.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Brain Cooling Treatment (Experimental): Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, during which they will wear a Welkins Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability. This brain cooling treatment will occur 5 days per week for 4 total weeks. Brain cooling treatment participants will also continue with their normally prescribed concussion recovery protocol as outlined by their outside clinicians.
  Interventions: Device: Brain Cooling
- Control (No Intervention): Control participants will maintain their normally prescribed concussion recovery protocol as outlined by their outside clinicians.

INTERVENTIONS:
Device: Brain Cooling — Brain cooling consists of a 30-minute seated period, in a dimly lit, quiet room, during which they will wear a Welkins Arctic Cooling Cap V1.30, set at a temperature of 33.0 degrees Fahrenheit. Participants will be asked to remain awake, refrain from observing a screen, and relax to the best of their ability. This brain cooling treatment will occur 5 days per week for 4 total weeks.
  Arms: Brain Cooling Treatment

SUMMARY:
This research is being done to examine the benefits of a 28 day head cooling intervention on cognition, inflammation of the brain, sleep quality, menstrual symptom interaction, and mood in acutely concussed females. Brain cooling has been shown to cause temporary symptom relief after traumatic brain injury, but its implications for decreasing timeline of full concussion recovery, particularly in females during periods of confounding neuropsychological menstrual symptoms, remains unexplored.

DETAILED DESCRIPTION:
Concussions are a form of mild traumatic brain injury (mTBI) that can lead to prolonged physical, cognitive, emotional, neuroinflammatory symptoms. An increase in IL-6 levels is seen due to neuroinflammation following mTBI. Following a concussion, females are more likely to experience sleep disturbances. This can impact the number of headaches and mood changes they experience. Emerging evidence suggests that hormonal fluctuations across the menstrual cycle may influence concussion recovery and symptoms specifically in the luteal phase.

Head cooling, or localized cranial hypothermia, has been explored as a therapeutic intervention to reduce neuroinflammation and cerebral metabolic demands following brain injury. Head cooling has been shown to reduce post-concussion symptoms recovery time and lessen the severity of symptoms like sleep disruptions, mood changes, and cognitive dysfunctions as well as decrease intracranial pressure. Recent research from our lab has also demonstrated that selective head cooling decreases depression symptoms and increases alpha wave power (measured via EEG). The gap that exists in the research is the effect that head cooling could have to help mitigate concussion symptoms specifically during the luteal phase of the menstrual cycle.

Thirty-two females, aged 18-27, will participate in this study (N=16 with acute concussion, N=16 healthy controls). Both sample groups will be randomly separated into placebo and head cooling intervention groups. The study will last the length of one pre-standardized menstrual cycle (28 days). The intervention group will receive 30-minute head cooling treatment, 5 days per week (Monday-Friday), while the placebo group will be instructed to continue normal daily activities without intervention. Participants will be asked to provide a blood sample on Day 1 and Day 28, which will be analyzed for serum concentration of Interluken-6 (IL-6), a neuroinflammatory biomarker. Also, on Day 1 and Day 28, participants will complete a brief cognitive testing battery that includes: the Psychomotor Vigilance Task (PVT), the Dual 2-Back, and the Stroop Task; as well as a brief psychological battery that includes: Beck's Depression Inventory-Fast Screen (BDI-fs), Hamilton Anxiety Rating Scale (HAM-A), and the Penn State Worry Questionnaire (PSWQ). Over the 28-day study timeline, participants will be asked to record their daily sleep using the free app, Consensus Sleep Diary (CSD) and record their daily menstrual cycle and symptoms using the free app, Clue, and record their daily concussion symptoms using a de-identified Qualtrics survey format Post-Concussion Symptom Scale (PCSS).

Visit 1 will occur on Day 1 of the study. Participants will be instructed to refrain from food, water, or brushing teeth for at least 30 minutes prior to their visit. At this time, the participants will be randomly assigned to the control or intervention group.

Participants will be asked to provide a blood sample, drawn by a registered nurse. This method requires the participants to have 5.0 mL of blood drawn. Samples will then be immediately stored in a marked freezer unit.

Next, the participants will be asked to complete a written history and demographics form, as well as the following mental health questionnaires: Beck's Depression Inventory-Fast Screen (BDI-fs), Hamilton Anxiety Rating Scale (HAM-A), and the Penn State Worry Questionnaire (PSWQ). After this, the subject will complete a computer-based cognitive testing battery that includes: the Psychomotor Vigilance Task (PVT), the Dual 2-Back, and the Stroop Task. These actions will only be completed out at the first visit (visit 1) and at the last visit (visit 2 for the control group, or visit 20 for the intervention group).

The subjects will also complete the Post-Concussion Symptom Scale (PCSS) during their first visit and will continue to do so daily until the last visit via a de-identified Qualtrics survey. On this daily survey participants will provide their given participant identification number, but not their name or any identifiable information.

The participant will then be informed about the Consensus Sleep Diary (CSD) app and the Clue app. They will create a de-identified account for each, which will be accessible by the study team for data collection purposes. Participants may download the application to their device or so use a personal computer so to access the applications and track their daily sleep and menstrual cycle & symptoms.

Participants assigned to the control group will be finished with Visit 1 at this time. Participants in the head cooling condition (intervention group) will undergo a 30-minute session while seated in a quiet, dimly lit room, listening to soothing natural sounds, wearing a Welkins Arctic Cooling Cap V1.30. The cap will be applied at room temperature and positioned on the top of the head, secured with adjustable Velcro straps; it does not include a chin strap. A coolant line connects the cap to the cooling system, which, when activated, circulates chilled coolant through the cap. The temperature of the cap will decrease from room temperature to 33.0°F over approximately 2-3 minutes. The cap remains dry and does not produce condensation during use. Pilot testing has shown that the cap is generally comfortable, but if a participant reports any discomfort, the cap will be immediately removed and adjusted. Sessions can also be ended at the participant's request. Participants will be instructed to remain awake, avoid looking at screens, and relax as much as possible.

The total duration of the first visit will last approximately 45 minutes for the control group and 75 minutes for the intervention group.

Visit 2 -19; the intervention group will come in everyday Monday-Friday for 30 minutes of head cooling (as explained above). That is, 20 total visits, over a 28 day period.

The control group will proceed with normal daily life during this time. The control group's next visit, which will be their Visit 2 and final visit, will occur at the same time as the intervention group's final visit. That is, 28 day (4 weeks), or one standard menstrual cycle, after Visit 1.

Thus, Visit 2 for control will be the same as visit 20 for the intervention group, and will occur 28 days after Visit 1. This visit will be the same as Visit 1 for both groups, however no head cooling will be administered to either group on this day. Thus, this final visit will last approximately 25 minutes for everyone.

ELIGIBILITY:
Inclusion Criteria:

1. Require that any participant is 18-27 years old
2. Require that participants be English speakers
3. Require that participants are females
4. Require that persons be able to provide consent for themselves

Exclusion Criteria:

1. Exclude persons under 18 years old or over 27 years old
2. Exclude persons taking anti-inflammatory drugs (both prescription and OTC), or those who will have taken them within 24 hours prior to Visit 1
3. Exclude smokers and former smokers, as defined by CDC. (Anyone who smokes daily or who has smoked at least 100 cigarettes in their lifetime)
4. Those with scalp infections, sun burns, skin cancers, and/or prior surgical scars should not participate
5. Those with presence of an active infection (including a dental infection)
6. Exclude persons who have migraines
7. Exclude persons taking mood stabilizer medications
8. Exclude persons who have consumed alcohol within 48 hours prior to study participation.
9. Exclude persons who are males

Ages: 18 Years to 27 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Beck's Depression Inventory-Fast Screen | The metrics will be assessed on pre-intervention (Day 1) and post-intervention (Day 28).
  The Beck's Depression Inventory-Fast Screen is a 13-item subjective report of depression symptoms.
HAM-A | The metrics will be assessed pre-intervention (Day 1) and post-intervention (Day 28).
  the HAM-A is a 14-item subjective report of anxiety symptoms.
The Penn State Worry Questionnaire | The metrics will be assessed pre-intervention (Day 1) and post-intervention (Day 28).
  The Penn State Worry Questionnaire is a 16-item subjective report of perceived worry.
Psychomotor Vigilance Task (PVT) | The metrics will be assessed pre-intervention (Day 1) and post-intervention (Day 28).
  The PVT is a very brief (<1 min) test to assess reaction time and sustained attention.
Dual 2-back Test | The metrics will be assessed pre-intervention (Day 1) and post-intervention (Day 28).
  The Dual 2-back Test is a 72 second measure of working memory.
Stroop Task | The metrics will be assessed pre-intervention (Day 1) and post-intervention (Day 28).
  The Stroop task is a brief measure of selective attention, processing speed, and executive function

SECONDARY OUTCOMES:
Consensus Sleep Diary (CSD) | CSD will be recorded daily throughout the intervention (from Day 1 to Day 28).
  The CSD is a remote application that allows for description and tracking of metrics related to sleep quantity and quality.
Clue App | Clue entries will be recorded daily throughout the intervention (from Day 1 to Day 28).
  The Clue App is a qualitative journaling tool for recording menstrual cycle timeline and symptom severity.
Post-Concussion Symptom Scale (PCSS) | PCSS will be recorded daily throughout the intervention (from Day 1 to Day 28).
  The PCSS is a 21 item concussion symptom self-scoring measure. Each item ranks a different concussion symptom category on a 0-6 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Recreation Building, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Congeni J, Murray T, Kline P, Bouhenni R, Morgan D, Liebig C, Lesak A, McNinch NL. Preliminary Safety and Efficacy of Head and Neck Cooling Therapy After Concussion in Adolescent Athletes: A Randomized Pilot Trial. Clin J Sport Med. 2022 Jul 1;32(4):341-347. doi: 10.1097/JSM.0000000000000916. Epub 2021 Mar 10. PMID 34009790
- [Background] Deng H, Han HS, Cheng D, Sun GH, Yenari MA. Mild hypothermia inhibits inflammation after experimental stroke and brain inflammation. Stroke. 2003 Oct;34(10):2495-501. doi: 10.1161/01.STR.0000091269.67384.E7. Epub 2003 Sep 11. PMID 12970518
- [Background] Leung LY, Cardiff K, Yang X, Srambical Wilfred B, Gilsdorf J, Shear D. Selective Brain Cooling Reduces Motor Deficits Induced by Combined Traumatic Brain Injury, Hypoxemia and Hemorrhagic Shock. Front Neurol. 2018 Aug 3;9:612. doi: 10.3389/fneur.2018.00612. eCollection 2018. PMID 30123177
- [Background] Westermaier T, Nickl R, Koehler S, Fricke P, Stetter C, Rueckriegel SM, Ernestus RI. Selective Brain Cooling after Traumatic Brain Injury: Effects of Three Different Cooling Methods-Case Report. J Neurol Surg A Cent Eur Neurosurg. 2017 Jul;78(4):397-402. doi: 10.1055/s-0036-1596057. Epub 2016 Dec 30. PMID 28038481
- [Background] Tan XR, Stephenson MC, Alhadad SB, Loh KWZ, Soong TW, Lee JKW, Low ICC. Elevated brain temperature under severe heat exposure impairs cortical motor activity and executive function. J Sport Health Sci. 2024 Mar;13(2):233-244. doi: 10.1016/j.jshs.2023.09.001. Epub 2023 Sep 9. PMID 37678507
- [Background] Walter A, Finelli K, Bai X, Johnson B, Neuberger T, Seidenberg P, Bream T, Hallett M, Slobounov S. Neurobiological effect of selective brain cooling after concussive injury. Brain Imaging Behav. 2018 Jun;12(3):891-900. doi: 10.1007/s11682-017-9755-2. PMID 28712093
- See also: publication from the Journal of Cerebral Blood Flow Metabolism describing use of this product in the methods — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9580175/